CLINICAL TRIAL: NCT06170450
Title: CYclic Versus Continuous Sacral Modulation for LowEr Urinary Tract Symptoms: a Prospective Randomized Controlled Trial (CYCLE Trial)
Brief Title: Cyclic Versus Continuous Sacral Neuromodulation for LUTS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Northwestern University (Other); University of Louisville (Other); Metro Health, Michigan (Other)
Responsible Party: Principal Investigator, David Sheyn, Physician, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY20231521
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Overactive Bladder Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cyclic SNM (Experimental): Programming of the SNM device will occur as per standard protocol in discussion between patient and SNM representative. The intervention will be to set the device to cycling stimulation program mode.
  Interventions: Device: Cyclic SNM
- Continuous SNM (Active Comparator): Programming of the SNM device will occur as per standard protocol in discussion between patient and SNM representative. The intervention will be to set the device to continuous stimulation programming (SNM is continuously stimulating without "off" periods)
  Interventions: Device: Continuous SNM

INTERVENTIONS:
Device: Cyclic SNM — SNM cycling: 8 hours on, 16 hours off
  Arms: Cyclic SNM
Device: Continuous SNM — Continuous SNM: on continuously, no 'off' period
  Arms: Continuous SNM

SUMMARY:
This will be a prospective, randomized-controlled multi-site trial comparing cyclic versus continuous sacral neuromodulation (SNM) for OAB.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is characterized by urinary frequency, urgency, incontinence, and nocturia in the absence of other pathology. AUA guidelines recommend trial of sacral neuromodulation (SNM) for patients with refractory OAB who have failed treatment with behavioral modification and medication. SNM settings are typically selected based on discussion between the patient and device representative. There is a paucity of rigorous data assessing optimal SNM stimulation programming for symptomatic improvement.

This will be a prospective, randomized-controlled multi-site trial comparing cyclic versus continuous sacral neuromodulation (SNM) in patients undergoing SNM for OAB.

Patients > age 18 with a diagnosis of refractory OAB being scheduled for a trial of SNM (either stage I lead/temporary battery placement or office peripheral nerve evaluation) will be approached by study personnel during their clinic visit or by a phone call to determine if they are interested in participating in the programming study.

Patients interested in participating will provide written informed consent. After informed consent is obtained, a baseline evaluation will be performed. This includes history, 3-day voiding diary (# voiding episodes, # nocturia episodes, # urge incontinence episodes/24h), urinalysis, urine culture (if indicated), post void residuals, and symptom assessments using questionnaires.

Only those with successful trial and eligible/ interested in permanent SNM placement will participate in this trial. Randomization will occur after stage 2/ full permanent implantation when the neuromodulator is being programmed in the recovery room. Patients will be randomly assigned to either continuous stimulation or cyclic stimulation.

Patients will then be followed with clinical evaluation and questionnaires repeated at 1 month, 6 months, 12 months, 3 years, and 5 years post-op.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Female
* English Speaking
* Diagnosis of urinary urge incontinence or overactive bladder
* Meet criteria for and are planning permanent SNM (ie. successful stage I or office PNE trial of SNM with 50% or more reduction in UUI episodes)
* Willing and able to complete all study related items

Exclusion Criteria:

* Patients less than 18 years of age
* Unable to provide consent
* Non-English speaking
* Relevant neurologic diseases (multiple sclerosis, Parkinson Disease, myasthenia gravis, - - - Charcot-Marie-Tooth disease, complete spinal cord injury)
* Current or prior bladder malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Change in ICIQ-OAB-QoL score | Baseline, 12 months post-operatively
  ICIQ-OABqol is a 28 question patient-completed survey evaluating quality of life (QoL) in patients with overactive bladder.

SECONDARY OUTCOMES:
Change in ICIQ-OAB-QoL score | Baseline, 1 month, 6 months, 12 months, 3 years, 5 years post-operatively
  ICIQ-OABqol is a 28 question patient-completed survey evaluating quality of life (QoL) in patients with overactive bladder.
Change in OAB-q SF | Baseline, 1 month, 6 months, 12 months, 3 years, 5 years post-operatively
  OAB-q SF is a 19 question patient-completed survey evaluating symptom bother and quality of life in patients with overactive bladder.
Change in Overactive Bladder Symptom Score (OABSS) | Baseline, 1 month, 6 months, 12 months, 3 years, 5 years post-operatively
  The Overactive Bladder Symptom Score (OABSS) is a 4 question validated symptom assessment tool for patients with OAB and assesses number of episodes of frequency, nocturia, urgency, and urge incontinence.
Change in Incontinence Impact Questionnaire SF (IIQ-7) | Baseline, 1 month, 6 months, 12 months, 3 years, 5 years post-operatively
  Incontinence Impact Questionnaire SF (IIQ-7) is a 7-item validated questionnaire that assesses urinary symptoms, the symptom bother, and the impact the bother has on patients' quality of life using a 4-point bother scale.
Urinary Distress Inventory SF (UDI-6) | Baseline, 1 month, 6 months, 12 months, 3 years, 5 years post-operatively
  Urinary Distress Inventory SF (UDI-6) is a 6 item validated questionnaire that assesses urinary symptoms, the symptom bother, and the impact the bother has on patients' quality of life using a 4-point bother scale.
Patient Global Impression of Severity (PGI-S) | Baseline, 1 month, 6 months, 12 months, 3 years, 5 years post-operatively
  Patient Global Impression of Severity (PGI-S) is a 1-item scale designed to assess for disease severity.
Patient Global Impression of Improvement (PGI-I) | Baseline, 1 month, 6 months, 12 months, 3 years, 5 years post-operatively
  Patient Global Impression of Improvement (PGI-I) is a 1-item scale designed to assess symptom improvement.
Overactive Bladder Satisfaction of Treatment Questionnaire | Baseline, 1 month, 6 months, 12 months, 3 years, 5 years post-operatively
  Change in Overactive Bladder Satisfaction of Treatment Questionnaire (OAB-SAT-q) is an 11-item validated questionnaire that assesses patients' satisfaction with their OAB treatment within a clinical setting from baseline.
Change in voiding frequency (# of voiding episodes in 24 hours) | Baseline, 1 month, 6 months, 12 months, 3 years, 5 years post-operatively
  Patients will use 3 days bladder diaries to track # of voids during the day, # of voids during the night, urgency episodes, and urge incontinence episodes. Daily voiding frequency will be the average # of voids per 24h averaged over 3 day bladder diary.
Change in nocturia episodes | Baseline, 1 month, 6 months, 12 months, 3 years, 5 years post-operatively
  Patients will use 3 days bladder diaries to track # of voids during the day, # of voids during the night, urgency episodes, and urge incontinence episodes. Nocturia episodes will be the average # of voids overnight per day averaged over 3 day bladder diary.
Change in urgency episodes | Baseline, 1 month, 6 months, 12 months, 3 years, 5 years post-operatively
  Patients will use 3 days bladder diaries to track # of voids during the day, # of voids during the night, urgency episodes, and urge incontinence episodes. Urgency episodes will be the average # of urgency episodes per 24h averaged over 3 day bladder diary.
Change in urinary urge incontinence episodes | Baseline, 1 month, 6 months, 12 months, 3 years, 5 years post-operatively
  Patients will use 3 days bladder diaries to track # of voids during the day, # of voids during the night, urgency episodes, and urge incontinence episodes. Urinary urge incontinence episodes will be the average # of urinary urge incontinence episodes per 24h averaged over 3 day bladder diary.

CONTACTS AND LOCATIONS:
Overall Officials: David Sheyn, MD, Principal Investigator — UH Hospitals Cleveland Medical Center
Locations (3):
- United States (3):
  - University of Louisville, Louisville, Kentucky
  - University Hospitals, Cleveland, Ohio
  - MetroHealth, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data will be shared with co-collaborators at Northwestern University (PI: Carol E. Bretschneider) and University of Louisville (PI: Ankita Gupta)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available during study recruitment and monitoring. When study has concluded, data will no longer be available.
Access Criteria: Available to only (IRB approved) members of study team through secure RedCap